CLINICAL TRIAL: NCT06560320
Title: The Effect of Using Virtual Reality Goggles on Fear and Pain Level During Vaccination in Children: A Randomized Controlled Study
Brief Title: Effect of Using Virtual Reality Goggles on Fear and Pain Level During Vaccination in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burdur Mehmet Akif Ersoy University (Other)
Responsible Party: Principal Investigator, Selda Ateş Beşirik, Principal Investigator, Burdur Mehmet Akif Ersoy University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GO 2024/176
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Fear of Pain; Fear; Virtual Reality; Pain; Vaccination; Children
Keywords: fear; Pain; Virtual Reality; Vaccination; Child; Children
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: This prospective, randomised controlled study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality Glasses Group (Experimental): Virtual Reality (VR) Glasses were introduced to the children pre-procedure. The children were made to watch a video with VR glasses before starting the application and it continued until the end of vaccination procedure.
  Interventions: Behavioral: Virtual Reality Glasses
- Control group (No Intervention): In this group, children received routine vaccination procedure.

INTERVENTIONS:
Behavioral: Virtual Reality Glasses — Virtual Reality(VR) Glasses were introduced to the children pre-procedure. The children were made to watch a video with VR glasses before starting the application and it continued until the end of the vaccination procedure.
  Arms: Virtual Reality Glasses Group

SUMMARY:
The study was designed as a randomized controlled experimental research with the purpose of determining the effect of distraction by using Virtual Reality Glasses reducing fear and pain during routine vaccination in children.

DETAILED DESCRIPTION:
In the literature, it is stated that nurses should use pharmacological and non-pharmacological methods in pain and anxiety management in painful procedures. Evidence-based studies are needed to show the effectiveness of non-pharmacological methods in reducing pain during invasive procedures and to investigate the effects of easy-to-apply methods on pain. In light of this information, this study aimed to examine the effect of distraction by using Virtual Reality Glasses in reducing fear and pain during routine vaccination in children.

This study is a prospective, randomized and controlled trial. Children aged 48 months who required routine vaccination were divided into two groups; Virtual Reality Glasses and Control. Data were obtained through face-to-face interviews with the children, their parents, and the observer before and after the procedure. The children's anxiety levels were also assessed using the Children's Fear Scale. The children's pain levels were assessed and reported by the parents and observers and the children themselves who selfreported using Wong-Baker FACES.

The study population consisted of the children's during routine vaccination in children aged 48 months. Sample of the study consisted of a total of 64 children who met the sample selection criteria and were selected via randomization method.

Children were randomized into two groups: Virtual Reality Glasses group (n= 32) and Control group (n= 32). Data were collected using the Interview and Observation Form, Children's Fear Scale, and Wong-Baker FACES Pain Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

* Children the ages of 48 months,
* Volunteering of the child and parent to participate in the study,
* Healthy children,
* Vaccination should be done by the same nurse,

Exclusion Criteria:

* The child has any acute or chronic disease,
* The child has a mental disability, vision, speech or communication problems,
* The parent has hearing, vision or verbal communication difficulties,
* The child used analgesics in the last 6 hours,
* Infection, disruption of skin integrity and rash in the area where the application will be made,
* Exclusion criteria were that the parent or child wanted to leave the study at any point.

Ages: 48 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Children's Fear Scale | Through painful procedure completion, an average of 10 minutes
  CFS is used for measuring the child's anxiety level. CFS is a scale which makes an evaluation from 0 to 4 consisting of five facial expressions drawn to show expressions that vary from neutral expression (0=no anxiety) to scared face (4=severe anxiety).
Wong-Baker FACES Pain Rating Scale | Through painful procedure completion, an average of 10 minutes
  In the study, pain level evaluations, the children's self-evaluations, parents' evaluations and the researcher's evaluations were carried out using the WB-FACES scale. This scale was developed by Donna Wong and Connie Morain Baker in 1988. The scale is graded between 0-10 points. A smiling face on the far left symbolizes "no pain" (0 very happy/no pain) and the pain increases from left to right. On the other hand, a crying face on the far right symbolizes "unbearable pain" (10 'hurts worst'). As the numbers increase in this scoring system, facial expressions also change referring to an increase in pain levels.

CONTACTS AND LOCATIONS:
Overall Officials: Selda Ateş Beşirik, Principal Investigator — Burdur Mehmet Akif Ersoy University
Locations (1):
- Burdur Bucak, Burdur, Bucak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this study, after deidentification, will be shared with researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code